CLINICAL TRIAL: NCT02488135
Title: Management of Persistent Anterior Epistaxis Using Floseal Hemostatic Matrix vs. Traditional Nasal Packing: A Prospective Randomized Controlled Trial.
Brief Title: Management of Persistent Epistaxis Using Floseal Hemostatic Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6601059
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-11

CONDITIONS: Epistaxis
Keywords: Floseal® (Baxter, USA); epistaxis; nasal packing; persistent
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Floseal Hemostatic Matrix (Experimental): Patients will receive Floseal Hemostatic Matrix topically at the location of active bleeding. Floseal is a gel-like fibrin glue that is applied using a syringe and forms a hemostatic clot.
  Interventions: Device: Floseal Hemostatic Matrix
- Traditional Nasal Packing (Active Comparator): Patients will receive traditional nasal packing to try and abort bleeding. This includes either vaseline gauze or nasal merocels being inserted into the anterior nasal cavity using forceps. These expand upon contact with blood or liquid therefore creating a compression type hemostasis.
  Interventions: Procedure: Traditional Nasal Packing

INTERVENTIONS:
Device: Floseal Hemostatic Matrix — Floseal Hemostatic Matrix is a gel like fibrin glue used topically in the nasal cavity and applied with a syringe.
  Arms: Floseal Hemostatic Matrix
Procedure: Traditional Nasal Packing — Using either vaseline gauze or nasal merocels. These will be placed in the anterior nasal cavity using nasal speculum and forceps.
  Arms: Traditional Nasal Packing

SUMMARY:
Nosebleeds that persist even after adequate traditional nasal packing may require aggressive treatment strategies to stop bleeding. Currently these strategies include a surgical approach to cut off blood supply to the vessel that is bleeding. FloSeal Hemostatic matrix is a gel like medical therapy that is inserted into the nose and is engineered to stop bleeding in severe cases, possibly avoiding the need for surgery. In this study the investigators will randomize patients to either receive FloSeal Hemostatix matrix or traditional nasal packing as a treatment for severe nosebleeds. The main outcome will be whether the investigators are able to stop bleeding with FloSeal or traditional packing alone and whether additional measures are necessary to stop the bleeding. The investigators will also perform a patient comfort survey and cost analysis. Even if FloSeal has equal effectiveness in treating nosebleeds as traditional packing, if it is much more comfortable for patients then it may be the favourable treatment.

DETAILED DESCRIPTION:
Background: Epistaxis is the most common emergent consultation to otolaryngology-head & neck surgery (OHNS) and with 60% of the population having experienced an episode and 1.6 in 10,000 requiring hospitalization in their lifetime. In preliminary studies Floseal® (Baxter, USA) Hemostatic Matrix has shown efficacy in up to 80% of persistent anterior epistaxis. We sought to evaluate the clinical efficacy¬ and cost-effectiveness of Floseal® (Baxter, USA) compared to traditional nasal packing for persistent epistaxis.

Methods: A prospective, randomized controlled trial was conducted on all adult patients consulted to the OHNS service at the tertiary referral centers of the University of Alberta Hospital and Royal Alexandra Hospital for persistent epistaxis. Patients were randomized to the Floseal® (Baxter, USA) or traditional packing study arms. Our main clinical outcome measures were: 1) Hemostasis directly following treatment and at 48 hours post-treatment, and 2) self-reported patient comfort at 48 hours post-treatment. Further, trial data was used for a formal cost-effectiveness analysis to determine incremental cost-effectiveness ratio (ICER). Univariate sensitivity analysis and uncertainty analysis were performed.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18+ presenting with epistaxis that requires an ENT consult that had a first attempt at treatment by an emergency physician.

Exclusion Criteria:

* Patients will be excluded based on the presence of a hypo-coagulable state. Including patients actively taking anti-coagulant medications or other patients with either acquired or hereditary bleeding disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cote, MD, FRCS(C), Principal Investigator — Alberta Health services
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murray S, Mendez A, Hopkins A, El-Hakim H, Jeffery CC, Cote DWJ. Management of Persistent Epistaxis Using Floseal Hemostatic Matrix vs. traditional nasal packing: a prospective randomized control trial. J Otolaryngol Head Neck Surg. 2018 Jan 8;47(1):3. doi: 10.1186/s40463-017-0248-5. PMID 29310703

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Floseal Hemostatic Matrix | Traditional Nasal Packing
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Floseal Hemostatic Matrix: Floseal Hemostatic Matrix provided as treatment.
- Traditional Nasal Packing: Traditional nasal packing provided as treatment.
- Total: Total of all reporting groups
Arm/Group | Floseal Hemostatic Matrix | Traditional Nasal Packing | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Full Range); unit: years] | 58.95 [22 to 95] | 55.08 [18 to 86] | 57.02 [18 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 13 | 13 | 26
Charlson Comorbidity Index [Mean (Full Range); unit: units on a scale] — The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes.
  Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient.
  A score of zero indicates that no comorbidities were found. The higher the score (max: 24) , the more likely the predicted outcome will result in mortality or higher resource use.
  units on a scale | 2.31 [0 to 7] | 2.31 [0 to 5] | 2.31 [0 to 7]
Aspirin Use [Count of Participants; unit: Participants] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Initial Hemostasis
Description: Residents administering the treatments will empirically observe primary hemostasis. Any active bleeding requiring further intervention within 4 hours of treatment will be defined as failure of initial hemostasis.
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Floseal Hemostatic Matrix | Traditional Nasal Packing
Number analyzed (Participants) | 13 | 13
Participants | 10 | 11
Statistical Analysis 1: Comparison: Floseal Hemostatic Matrix vs Traditional Nasal Packing; Test type: Non-Inferiority — An a priori sample size was calculated using a non-inferiority limit (d) set at 25%, significance level (α) of 5% and power of 80%. We assumed that success in each group would be 93% based on the literature examining anterior nasal packing in ideal conditions and considering our selection criteria in the Floseal® (Baxter, USA) population. Attrition was assumed to be 0% due to the short duration of treatment. This yielded 26 participants with 13 patients in each study arm; p = 1.000, Fisher Exact

2. Secondary Outcome: Patient Pain Level
Description: Patients will be contacted 48 hours following treatment with either Floseal or traditional nasal packing and be asked to rate their pain on a 10-point "Visual Analog Pain Scale". They will rate their pain for: 1) the placement of the treatment, 2) the duration of the treatment AND 3) the removal of the treatment.
  Minimum: 0 (less pain) Maximum: 10 (more pain)
  Higher scores indicate more pain and lower scores indicate less pain.
Time Frame: 48 hours
Population: Patients that failed initial hemostasis were traditionally packed and therefore were not able to rate either treatment or removal of the product.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Floseal Hemostatic Matrix | Traditional Nasal Packing
Number analyzed (Participants) | 12 | 13
units on a scale
  Pain Score During Placement | 2.42 [0 to 8] | 7.77 [4 to 10]
  Pain Score During Treatment: number analyzed (Participants) | 9 | 13
  Pain Score During Treatment | 0.50 [0 to 3] | 4.46 [0 to 10]
  Pain Score During Removal: number analyzed (Participants) | 9 | 13
  Pain Score During Removal | 0 [0 to 0] | 3.85 [0 to 10]
Statistical Analysis 1: Comparison: Floseal Hemostatic Matrix vs Traditional Nasal Packing; Comparison between groups for pain during placement; Test type: Superiority; p = 0.0022, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Floseal Hemostatic Matrix vs Traditional Nasal Packing; Comparison between groups for pain during treatment; Test type: Superiority; p = 0.0007, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Floseal Hemostatic Matrix vs Traditional Nasal Packing; Comparison between scores for pain during removal; Test type: Superiority; p = 0.0021, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Floseal Hemostatic Matrix | Traditional Nasal Packing
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Lack of blinding to either patient or practitioner. 30 day follow-up limit on outcomes and adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-06-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT02488135/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT02488135/SAP_001.pdf
  • Informed Consent Form (2015-08-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT02488135/ICF_002.pdf